CLINICAL TRIAL: NCT01626222
Title: A Phase IIIB, Multi-Center, Open Label Study For Postmenopausal Women With Estrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer Treated With Everolimus (RAD001) in Combination With Exemestane: 4EVER - Efficacy, Safety, Health Economics, Translational Research
Brief Title: 4EVER - Efficacy, Safety, Health Economics, Translational Research of Postmenopausal Women With Estrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer
Acronym: MACS2096
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001JDE49
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Postmenopausal; Estrogen Receptor Positive; HER2 negative; Locally Advanced; Metastatic Breast Cancer; Everolimus (RAD001); Exemestane
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus & Exemestane (Experimental): This study will be performed in 300 postmenopausal women with hormone receptor positive locally advanced or metastatic breast cancer progressing following prior therapy with non-steroidal aromatase inhibitors (NSAI) as defined by: 1. Recurrence while on or after completion of an adjuvant treatment including Letrozole or Anastrozole, or 2. Progression while on or following the completion of Letrozole or Anastrozole treatment for locally advanced or metastatic breast cancer. Except for prior use of mTOR inhibitors, there are no restrictions as to the last anticancer treatment prior to enrollment. Patients must have documented evidence of recurrence or progression on last therapy prior to enrollment. Written informed consent must be obtained prior to any screening procedures. The investigator or designee must ensure that only patients who meet all the following inclusion and none of the exclusion criteria are offered enrollment in the study.
  Interventions: Drug: Exemestane; Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Exemestane — Exemestane is supplied by Novartis until Everolimus is commercially available for the study setting. Afterwards the investigator will prescribe Exemestane according to the individual label. Commercially available Exemestane will be supplied as tablets of 25 mg strength for oral administration. Complete guidelines for management and administration of Exemestane can be found in the package insert. Exemestane will be dosed starting on treatment Day 1. Patients will be instructed to take 1 tablet of 25 mg Exemestane orally. Package insert instructions should be followed. On the first day of each cycle, patients will receive an adequate drug supply (before commercial availability) or a prescription (after commercial availability) for self-administration at home. The investigator must emphasize compliance and will instruct the patient to take Exemestane exactly as prescribed.
Drug: Everolimus (RAD001) — Everolimus (RAD001) is supplied by Novartis until Everolimus is commercially available for the study setting. Afterwards the investigator will prescribe Everolimus according to the individual label. Everolimus is formulated as tablets of 10 and 5 mg strength for oral administration. All study medication will be packaged into blister packs. The blisters should be opened only at the time of administration, as the drugs are both hygroscopic and light sensitive. Everolimus will be dosed starting on treatment Day 1. Patients will be instructed to take 1 tablet × 10 mg Everolimus orally with a large glass of water once daily at the same time each day with or without food. On the first day of each cycle, patients will receive an adequate drug supply (before commercial availability) or a prescription (after commercial availability) for self-administration at home. The investigator must emphasize compliance and will instruct the patient to take Everolimus exactly as prescribed.

SUMMARY:
The present multi-center, open-label, single-arm study aims to evaluate the efficacy and safety, quality of life and health resources utilization in postmenopausal women with hormone receptor positive breast cancer progressing following prior therapy with non-steroidal aromatase inhibitors (NSAI) treated with the combination of Everolimus and Exemestane.

DETAILED DESCRIPTION:
In light of the need for new treatment options for postmenopausal, hormone receptor positive, HER2 negative women after failure of prior non-steroidal aromatase inhibitor (NSAI) therapy, the BOLERO-2 trial was performed and demonstrated significant efficacy of the combinatorial treatment of Everolimus and Exemestane compared to an Exemestane monotherapy in this setting.

In this randomized, double blind, placebo-controlled trial a statistically significant improvement in progression-free survival (PFS) by adding Everolimus to exemestane versus Exemestane alone was reported. Adding Everolimus determined a 2.4-fold prolongation in PFS from 3.2 up to 7.4 months and so lowered the risk of cancer progression by 56% for these women. These findings were confirmed by an independent assessment (4.1 vs. 11.0 months, risk reduction: 64%). The quality of life data shows positive trend in the Everolimus plus Exemestane treatment arm. (Baselga 2011, Hortobagyi 2011). Thus, the benefit of the combinatorial treatment versus Exemestane monotherapy was shown in a defined patient population under controlled conditions.

The primary objective of this trial to assess the Overall Response Rate (ORR) in postmenopausal women with hormone receptor positive breast cancer progressing following prior therapy with NSAIs treated with the combination of Everolimus and Exemestane. The secondary objectives include, Progression free survival (PFS), Overall survival (OS), Safety, Change in Quality of life scores over time, Health resource utilization. The exploratory objectives reflect scientific interest within the treatment of metastatic breast cancer and are to be modified, if applicable, according to the current scientific state of the art at the time of actual analysis. These include: the influence of age, performance status, cancer activity and inflammation on anxiety and depression; changes in serum bone-turnover biomarkers; Pharmacogenetics of Everolimus in patients with advanced breast cancer; presence and molecular characteristics of Circulating Tumor Cells; correlation of response to Exemestane/Everolimus with Proteomic analysis.

The present national, multi-center, open-label, single-arm study aims to evaluate the efficacy and safety, quality of life and health resources utilization of the combination of Everolimus and Exemestane in a broader patient population compared to BOLERO-2, i.e. without limitations as to the number of previous chemotherapy lines, the time point of progression after NSAI therapy, and the previous endocrine therapy as patients under Exemestane monotherapy may be enrolled. Since the combination was shown to significantly improve PFS in the previous BOLERO-2 trial, for ethical reasons no endocrine comparator drugs will be investigated in the present study, due to the low efficacy of Exemestane monotherapy (PFS 3.2 months).

ELIGIBILITY:
Main Inclusion criteria:

Metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy or any other non-systemic treatment.

Histological or cytological confirmation of estrogen receptor positive (ER+) and/or progesterone receptor positive (PgR+), human epidermal growth factor receptor 2 (HER2) negative breast cancer Postmenopausal women. Disease progression following prior therapy with non steroidal aromatase inhibitors (NSAI), defined as: Recurrence while on, or following completion of an adjuvant treatment with Letrozole or Anastrozole, or Progression while on or following completion of Letrozole or Anastrozole treatment for ABC/MBC.

Radiological evidence of recurrence or progression on last systemic therapy prior to enrollment.

Patients must have at least one lesion that can be accurately measured or bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease.

Written informed consent obtained before any screening procedure and according to local guidelines.

Other protocol defined inclusion criteria apply.

Main Exclusion criteria:

HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).

Patients with only non-measurable lesions other than bone metastasis (e.g. pleural effusion, ascites etc.).

Previous treatment with mTOR inhibitors or known hypersensitivity to mTOR inhibitors.

Symptomatic brain or other CNS metastases. Previously treated brain metastases are allowed provided the patient is free of symptoms, prior radiotherapy for brain metastasis was more than four weeks before enrollment and the dose of corticosteroids is low (i.e. ≤ 10 mg/d Prednisolone equivalent) and stable for at least two weeks prior to enrollment.

Patients with Hepatitis B or C or with a history of Hepatitis B or C. Patients unwilling to or unable to comply with the protocol. Other protocol defined exclusion criteria apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) after 24 weeks of treatment | 24 weeks
  The Overall response rate (ORR) is the proportion of patients with a best overall response of confirmed complete (CR) or partial (PR) response by Week 24. The best overall response is determined from the sequence of investigator overall lesion responses according to RECIST 1.1. To be assigned a best overall response of CR at least two determinations of CR at least 4 weeks apart before progression are required. To be assigned a best overall response of PR at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) are required.

SECONDARY OUTCOMES:
Progression free survival (PFS) after 48 weeks of treatment | 48 weeks
  Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Overall Response Rate (ORR) after 48 weeks of treatment | 48 weeks
  The ORR by Week 48 will be derived from the sequence of overall lesion responses as described for the primary efficacy variable. The ORR by Week 48 will be summarized using frequency tables presenting absolute and relative frequencies together with appropriate confidence intervals
Overall survival (OS) after 48 weeks of treatment | 48 weeks
  Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact. OS will be summarized using the Kaplan-Meier method.
Safety within 48 weeks of treatment | 48 weeks
  The assessment of safety will be based mainly on the frequency of adverse events and on the number of laboratory values that fall outside of pre-determined ranges. Other safety data (e.g. vital signs, and special tests) will be considered as appropriate. For all safety analyses, the safety set will be used.
Resource utilization | 48 weeks
  Data relating to Resource Utilization will be used for the purpose of economic evaluation, which will be carried out and reported as a separate activity.
  The study population receiving RAD001 plus Exemestane will be compared to alternative cohorts (e.g., purely endocrine treatment with Fulvestrant monotherapy, Exemestane monotherapy or chemotherapy, e.g. Capecitabine) using a Markov model. For each alternative therapy option, median PFS, OS and health-related quality of life will be determined by a systematic review of literature or databases.
Health-related quality of life | 48 weeks
  Health-related quality of life (HRQoL) will be assessed using the EORTC QLQ-C30 and BR23 questionnaires and the EuroQoL EQ-5D questionnaire. The HADS D questionnaire will be used to assess anxiety and depression. Scoring will follow the instructions of the respective manuals.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (69):
- Germany (69):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Amberg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bergisch Gladbach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Eutin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Plauen-Kauschwitz
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Rosenheim
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stralsund
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Weißenfels
  - Novartis Investigative Site, Wuppertal

REFERENCES:
- [Derived] Hadji P, Stoetzer O, Decker T, Kurbacher CM, Marme F, Schneeweiss A, Mundhenke C, Distelrath A, Fasching PA, Lux MP, Luftner D, Janni W, Muth M, Kreuzeder J, Quiering C, Grischke EM, Tesch H. The impact of mammalian target of rapamycin inhibition on bone health in postmenopausal women with hormone receptor-positive advanced breast cancer receiving everolimus plus exemestane in the phase IIIb 4EVER trial. J Bone Oncol. 2018 Oct 2;14:010-10. doi: 10.1016/j.jbo.2018.09.010. eCollection 2019 Feb. PMID 30515367
- [Derived] Tesch H, Stoetzer O, Decker T, Kurbacher CM, Marme F, Schneeweiss A, Mundhenke C, Distelrath A, Fasching PA, Lux MP, Luftner D, Hadji P, Janni W, Muth M, Kreuzeder J, Quiering C, Taran FA. Efficacy and safety of everolimus plus exemestane in postmenopausal women with hormone receptor-positive, human epidermal growth factor receptor 2-negative locally advanced or metastatic breast cancer: Results of the single-arm, phase IIIB 4EVER trial. Int J Cancer. 2019 Feb 15;144(4):877-885. doi: 10.1002/ijc.31738. Epub 2018 Oct 30. PMID 29992557